CLINICAL TRIAL: NCT00004760
Title: Study of Axial Mobility Exercises in Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Educational/Counseling/Training
Other Study IDs: 199/11694; DUMC-722955R2
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Neurologic and psychiatric disorders; Rare disease
MeSH Terms: conditions — Parkinson Disease; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Exercise

INTERVENTIONS:
Behavioral: Exercise

SUMMARY:
OBJECTIVES:

I. Compare the benefit of exercise versus usual care (no exercise) on impairments and functional limitations in patients with Parkinson disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Patients assigned to the Axial Mobility Exercise Program participate 3 times a week for 10 weeks. The program consists of individualized exercises specifically directed toward restoration of axial mobility in the context of functional tasks.

Patients assigned to the control group receive standard care (no exercise).

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Stage 2 or 3 Parkinson disease (Hoehn/Yahr scale) Able to ambulate independently Able to function independently in home Moderate rigidity No moderate or severe tremor --Prior/Concurrent Therapy-- Concurrent stable pharmacologic regimen required --Patient Characteristics-- Cardiovascular: No unstable angina Other: No psychiatric or medical contraindication to exercise, e.g., dementia, hip fracture; no other neurologic disorder, e.g., stroke, multiple sclerosis; resides within 30 miles of Duke University

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 1995-05; Study Completion 1997-12

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Schenkman, Study Chair — Duke University

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886